CLINICAL TRIAL: NCT01097213
Title: Collaboration on Alcohol Self Administration in Adolescents and Young Adults - Specific Aim 2: To Examine the Effect of Acute Alcohol Administration on Forebrain Disinhibition Using Functional Magnetic Resonance Imaging (fMRI)
Brief Title: Neural Mechanisms Underlying Alcohol Induced Disinhibition
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: U01 AA017900 SA2; U01AA017900 (NIH)
Record Dates: First submitted 2010-03-11; First posted 2010-04-01 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ethanol — Intravenous infusion of 6% ethanol in half-normal saline for approximately 1 hour: The dosage is controlled by a physiologically-based pharmacokinetic (PBPK) model of alcohol distribution and elimination, developed by O'Connor and his associates at the Indiana Alcohol Research Center (IARC) (Ramchandani et al, 1999). PBPK Parameters that determine the dosage and frequency of the infusion for a specific individual are estimated by means of morphometric variables (age, height, weight and gender).
Drug: Placebo - half-normal saline — Intravenous infusion of half-normal saline for approximately 1 hour: The dosage is equal to the infusion dosage estimated by the PBPK model of alcohol distribution and elimination (Ramchandani et al., 1999) for the drug - ethanol condition.

SUMMARY:
Forty 18-year-old social drinkers will be selected from the sample tested in specific aim 1 ("Prospective Assessment of Adolescent Drinking Trajectories With Computer-Assisted Self-administration of Ethanol (CASE)"; ClinicalTrials.gov identifier: NCT01063166). The functional magnetic resonance imaging blood-oxygen-level-dependent (fMRI BOLD) activity related to disinhibition measured with the Stop Signal task will be assessed during a continuous infusion of alcohol, clamping the arterial Breath Alcohol Concentration (aBAC) at 60 mg% for approximately one hour. It will be examined whether this fMRI BOLD activity is associated with the initial drinking trajectories and the alcohol consumption at age 18 and at age 20 identified in specific aim 1. Furthermore, fMRI will be used with the Taylor Aggression Paradigm to determine which brain areas mediate increased physical aggression during the same continuous infusion of alcohol as described above. All participants will undergo an alcohol and a placebo fMRI session.

ELIGIBILITY:
Inclusion Criteria:

* male and female Caucasian volunteers aged 18 years/0 months to 19 years/11 months;
* written informed consent by the subject;
* habitual social drinking during the two months preceding participation, defined by at least one drinking day in any two weeks-interval;
* at least one prior experience of alcohol intoxication
* being able to abstain from tobacco use for four hours without developing nicotine withdrawal symptoms;
* effective contraception in female participants;
* consenting to abstain from any illegal substance use for 2 weeks prior to participation;
* living within 15 km (9.5 miles) from downtown Dresden;
* sufficient information concerning alcohol use in both parents and in at least four second-degree relatives

Exclusion Criteria:

* prior medical treatment due to alcohol use;
* current or prior history of any serious disease, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, alcohol or drug dependence, but not alcohol abuse;
* current history of Axis-I psychiatric illness, including premenstrual dysphoric disorder;
* current or prior history of alcohol-induced flushing reactions;
* positive urine screen for cannabinoids, cocaine, amphetamines, opiates, or benzodiazepines;
* light or non-drinkers: averaging less than 2 standard drinks per week in the preceding two months;
* intention to become pregnant
* pregnancy or positive urine pregnancy screening or breast-feeding;
* any alcohol intake on the test day or the day before;
* use of medications known to interact with alcohol within 2 weeks of the study;
* positive hepatitis or HIV at screening, provided the subject consented to these tests
* any conditions posing safety issues with the fMRI scan, such as ferromagnetic implants, cardiac pacemakers or insulin pumps

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents living within 15 km (9.5 miles) from downtown Dresden
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | 2 years
  Alcohol consumption, as measured by a Timeline Followback Interview.

SECONDARY OUTCOMES:
Absolute perfusion levels assessed with arterial spin labeling | 1 week
Behavioural Stop Signal Reaction Time (SSRT) | 1 week
BOLD fMRI correlate of aggression | 1 week
Taylor aggression score | 1 week
BOLD fMRI correlate of disinhibition | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Michael N. Smolka, Prof. Dr., Principal Investigator — Technische Universitaet Dresden - - Faculty of Medicine Carl Gustav Carus - Department of Psychiatry and Psychotherapy; Ulrich S. Zimmermann, Dr., Principal Investigator — Universitaetsklinikum Carl Gustav Carus at the Technische Universitaet Dresden
Locations (1):
- Technische Universitaet Dresden - Dresden fMRT-Neuroimaging Center, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Gan G, Guevara A, Marxen M, Neumann M, Junger E, Kobiella A, Mennigen E, Pilhatsch M, Schwarz D, Zimmermann US, Smolka MN. Alcohol-induced impairment of inhibitory control is linked to attenuated brain responses in right fronto-temporal cortex. Biol Psychiatry. 2014 Nov 1;76(9):698-707. doi: 10.1016/j.biopsych.2013.12.017. Epub 2014 Jan 15. PMID 24560581